CLINICAL TRIAL: NCT02810132
Title: Effects of Metformin Treatment on Myocardial Efficiency in Patients With Heart Failure: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effects of Metformin Treatment on Myocardial Efficiency in Patients With Heart Failure
Acronym: METRONOME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Wiggers, Senior consultant, associate professor, PhD, DMSc, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-588
Record Dates: First submitted 2016-06-08; First posted 2016-06-22 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Drug: Metformin Target dose: 1000 mg x 2 (if eGFR 30-60 ml/min: 500 mg x 2) Other name: Glucophage XR 500
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — See above
  Other Names: Glucophage XR 500
  Arms: Metformin
Drug: Placebo — See above
  Arms: Placebo

SUMMARY:
The study evaluates the effects of metformin treatment on myocardial efficiency in heart failure patients. 36 patients will be randomized to three months of metformin or placebo treatment in addition to their regular therapy.

Hypothesis: Treatment with metformin in patients with heart failure has direct or indirect beneficial effects on left ventricular myocardial oxidative metabolism, myocardial efficiency and contractile function.

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a common disease and diabetes/insulin resistance are present in approximately 50 % of HF patients. Metformin is the most commonly prescribed oral anti-diabetic drug, and registry and experimental studies show beneficial effects of metformin in HF, but randomized trials are needed.

Objectives: To investigate if treatment with metformin in patients with HF has beneficial effects on myocardial efficiency,

Design: A randomized, double-blind, placebo-controlled, single-center design. 36 patients with systolic heart failure will be randomized to either metformin (N = 18) or placebo (N= 18) for 3 months.

Methods: Patients will undergo echocardiography at rest and during exercise along with [11C]-acetate PET.

Primary outcome parameter is changes in myocardial external efficiency from visit 1 to 3 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure uptitrated to recommended or maximally tolerated dose of ACE-I/ARB (unless contraindicated) and beta-blocker (unless contraindicated). If indicated, an aldosterone receptor antagonist should be given (unless contraindicated). An ICD and/or CRT should be implanted, if indicated. Patients with a CRT device should be treated for > 3 months.
* LVEF < 45%
* NYHA-class II, III or IV
* Relatively preserved renal function (eGFR > 30 ml/min)
* Ability to understand the written patient information and to give informed consent
* Negative urine-HCG for women of childbearing potential
* Patients must have insulin resistance, defined as 1 or more of the following criteria:

  1. HbA1c 5.5 - 6.4% (37 - 47 mmol/mol) within the last 12 months prior to enrolment
  2. Impaired fasting glucose (IFG): Fasting P-glucose 5.6 - 6.9 mmol/l within 12 months prior to enrolment (patient in stable condition)
  3. Impaired glucose tolerance (IGT) if OGTT has been performed at any time prior to enrolment: Fasting P-glucose < 7.0 mmol/l and 2 hour P-glucose 7.8 -11.0 mmol/l

Exclusion Criteria:

* Metformin treatment within the last 3 months
* Known allergy to metformin or major side effects to metformin treatment
* Acute myocardial infarction, unstable angina or revascularization < 3 months at the time of randomization
* Planned coronary revascularization
* Significant, uncorrected cardiac valve disease
* Cardiac arrest or life threatening ventricular arrhythmias within the last 3 months (unless treated with an ICD)
* Atrial fibrillation with poorly controlled ventricular rate at rest (> 100 beats/min)
* Hypertrophic or restrictive cardiomyopathy, infiltrative or storage myocardial disease, active myocarditis, or pericardial disease.
* Planned major surgery
* Female patients who are pregnant, nursing, or of childbearing potential while not practicing effective chemical contraceptive methods (i.e. oral, implanted, injectable, or transdermal contraceptive hormones; intrauterine device)
* Age < 18 years
* Current abuse of alcohol or drugs
* Cancer, with a life-expectancy of less than 2 years
* Stroke within the last 6 months
* Liver disease with P-ALAT >3 times upper normal limit (it is possible to repeat this measurement once within a month)
* Significant comorbidity or issue that makes the patient unsuitable for participation as judged by the investigator
* Participation in another study involving long-term medical intervention (participation in device studies is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Changes in LV myocardial efficiency | Baseline and 3 months
  LV myocardial efficiency is the ratio between stroke work and myocardial oxygen consumption, which are measured with echocardiography and [11C]-acetate PET.

SECONDARY OUTCOMES:
Left ventricular global longitudinal strain during peak exercise | Baseline and 3 months
Myocardial oxygen consumption | Baseline and 3 months
Myocardial perfusion at rest | Baseline and 3 months
LV myocardial function evaluated by LVEF and diastolic function | Baseline and 3 months
LV mass | Baseline and 3 months
6 minute walking distance | Baseline and 3 months
Changes in body composition | Baseline and 3 months
  Measured by bioelectrical impedance analysis (BIA)
Maximum oxygen consumption | Baseline and 3 months
Degree of insulin resistance | Baseline and 3 months
Minnesota living with heart failure questionnaire | Baseline and 3 months
NT-proBNP | Baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Palle Juul-Jensens Boulevard 99, Aarhus N, Denmark

REFERENCES:
- [Derived] Larsen AH, Wiggers H, Dollerup OL, Jespersen NR, Hansson NH, Frokiaer J, Brosen K, Norrelund H, Botker HE, Moller N, Jessen N. Metformin Lowers Body Weight But Fails to Increase Insulin Sensitivity in Chronic Heart Failure Patients without Diabetes: a Randomized, Double-Blind, Placebo-Controlled Study. Cardiovasc Drugs Ther. 2021 Jun;35(3):491-503. doi: 10.1007/s10557-020-07050-5. Epub 2020 Aug 8. PMID 32770520